CLINICAL TRIAL: NCT03416712
Title: Transforming Care and Payment Priorities for Vulnerable Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Michelle Lopez, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: H-38428
Record Dates: First submitted 2017-10-03; First posted 2018-01-31 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Social Stress
Keywords: Social Determinants of Health
MeSH Terms: interventions — Health Resources

STUDY DESIGN:
Intervention Model Description: Quantify unmet socioeconomic determinants of health (SDH) needs using a screening tool in the inpatient settings at Texas Children's Hospital (TCH). Screen will assess educational attainment, employment, literacy, language skills, substance dependence, childcare and child behavior, mental health, domestic violence, housing insecurity and conditions, medical insurance, access to primary care, transportation to medical appointments, ability to pay for prescriptions, legal issues and immigration services. 2. Increase vulnerable family enrollment in community resources to decrease unmet psychosocial and economic needs in the study population 3. Evaluate impact of this intervention on health outcome indicators and hospital resource utilization (body mass index (BMI), return visit to ED, hospital readmission, and parent's perception of child's health).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): To obtain baseline socioeconomic data on all children (intervention and control), study participants will utilize the Children's HealthWatch Survey (www.childrenshealthwatch.org), which is a standardized, validated survey designed to collect demographics and information on child health and development, parental health, and socioeconomic factors income, education level, financial literacy, childcare, and government assistance).
  The control group will not complete the WE CARE HOUSTON survey and will not receive any referrals to community resources from the study team at the time of enrollment (they may be referred to resources by their medical/clinical team as per standard of care during their hospitalization at Texas Children's Hospital). The study investigators will offer control participants information on community resources at the end of the study. Study participants will be called for a 6 month follow up structure telephone survey.
- Intervention (Experimental): The intervention group will complete a short survey called the WE CARE HOUSTON survey. The WE CARE HOUSTON survey has been designed to quickly assess patient need for local services that address the social determinants of health. The WE CARE HOUSTON survey will be administered on paper or verbally if family is not able to read. Based on the parent's responses to the screening survey, the study investigators will use an algorithm to direct families to appropriate services and community resources. Families who screen positive for social needs will receive a handout on resources. For the families that screen positive for depression/ mental health needs, domestic violence, or alcohol and drug abuse, the study investigators will notify the medical/clinical team and recommend an inpatient social work prior to discharge. Intervention participants will be called 1 week-2 months after enrollment to follow up on resources and will be called for a 6 month follow up structured telephone survey.
  Interventions: Other: Screening survey and accompanying handout for resources

INTERVENTIONS:
Other: Screening survey and accompanying handout for resources — Intervention group will be completing a survey of social determinants of health and providing resources based on caregiver responses.
  Other Names: Addressing social needs
  Arms: Intervention

SUMMARY:
This will be a randomized control trial of 800 children admitted to the Pediatric Hospital Medicine service at Texas Children's Hospital. Each eligible participant will give informed consent prior to enrollment. Study participants will be randomized into an intervention (400 participants) or control group (400 participants). The intervention group will receive a survey (WE CARE HOUSTON) that has been designed to assess family need for community resources that address the SDH (such as food insecurity, housing insecurity, etc.). The intervention group will receive referrals to community resources based on their responses to the WE CARE HOUSTON survey.

DETAILED DESCRIPTION:
This will be a randomized control trial of 800 children admitted to the Pediatric Hospital Medicine service at Texas Children's Hospital. Each eligible participant will give informed consent prior to enrollment.

Study participants will be randomized into an intervention (400 participants) or control group (400 participants). The intervention group will receive a survey (WE CARE HOUSTON) that has been designed to assess family need for community resources that address the SDH (such as food insecurity, housing insecurity, etc.). The intervention group will receive referrals to community resources based on their responses to the WE CARE HOUSTON survey. The intervention group will receive a phone call within 3 months of discharge to ask if they have had trouble following up with resources.

Both the intervention and the control groups will be followed for 6 months. Study investigators will obtain outcome data through structured telephone interviews at 6 months and also through medical record review.

This research has been designed to test our hypotheses:

1. The use of the WE CARE HOUSTON screening tool and subsequent referral to community resources will result in increased family participation in community resources that address the SDH; i.e. we believe that the intervention group will enroll in more community resources than the control group over the 6 month study period.
2. The use of the WE CARE HOUSTON screening tool and subsequent referral to community resources will result in improved health outcomes, i.e. children in the intervention group will have fewer emergency department visits, fewer readmissions, improved BMI and improved parent perception of child's health during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Children admitted to pediatric hospital medicine service

Exclusion Criteria:

* Children in child protective service custody
* Children residing outside of the greater Houston area

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 430 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Enrollment (yes/no) in social determinant of health resources based on answer to questionnaire | 6 months after study enrollment
  We will assess whether study participants followed up with the resources provided and were able to enroll in needed resources with follow up phone call.

SECONDARY OUTCOMES:
Decreased emergency department revisits and hospital readmissions | 6 months after study enrollment
  We will assess whether children in the intervention group will have fewer quantity of all cause emergency department visits, fewer quantity of hospital readmissions on chart review.
Improved parental perception of child's health | study enrollment to 6 months after enrollment
  We will compare caregiver's baseline and 6 month self-rating of their child's health in categories of "excellent", "good", "fair" or "poor".
Child's immunization status | 6 months after study enrollment
  Self report of compliance with vaccinations by parents on follow up survey
Child's growth | 6 months after study enrollment
  Weight and height will be combined to report BMI in kg/m^2. If height is unavailable, weight will be used and reported in kilograms.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Lopez, MD, MPH, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garg A, Toy S, Tripodis Y, Silverstein M, Freeman E. Addressing social determinants of health at well child care visits: a cluster RCT. Pediatrics. 2015 Feb;135(2):e296-304. doi: 10.1542/peds.2014-2888. Epub 2015 Jan 5. PMID 25560448
- [Background] Garg A, Butz AM, Dworkin PH, Lewis RA, Thompson RE, Serwint JR. Improving the management of family psychosocial problems at low-income children's well-child care visits: the WE CARE Project. Pediatrics. 2007 Sep;120(3):547-58. doi: 10.1542/peds.2007-0398. PMID 17766528
- [Background] Garg A, Butz AM, Dworkin PH, Lewis RA, Serwint JR. Screening for basic social needs at a medical home for low-income children. Clin Pediatr (Phila). 2009 Jan;48(1):32-6. doi: 10.1177/0009922808320602. Epub 2008 Jun 19. PMID 18566347
- [Derived] Lopez MA, Yu X, Hetrick R, Raman S, Lee J, Hall J, Tran K, Vonasek B, Garg A, Raphael J, Bocchini C. Social Needs Screening in Hospitalized Pediatric Patients: A Randomized Controlled Trial. Hosp Pediatr. 2023 Feb 1;13(2):95-114. doi: 10.1542/hpeds.2022-006815. PMID 36594231